CLINICAL TRIAL: NCT06681272
Title: Prediction of Chronic Pain in Cardiac Surgery: Evaluation by Algocartography
Brief Title: Prediction of Chronic Pain in Cardiac Surgery: Evaluation by Algocartography Predict-ALGOCARTE
Acronym: Predict-ALGOCA
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0457; 2024-A01249-38 (Other: ID-RCB)
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sternotomy Closure,Open Heart Surgery; Cardiac Surgery; Chronic Pain Post-Procedural
Keywords: Chronic pain prediction; cardiac surgery; algocartography; area of hyperalgesia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients undergoing scheduled sternotomy cardiac surgery: Cohort, cardiac surgery patients who develop chronic pain Chronic post-surgical pain is defined as pain localized to the surgical site, with no other attributable cause, that persists for more than three months after surgery and has an impact on quality of life.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — sleep quality assessment using the PROMIS (Patient-Reported Outcomes Measurement Information System) item Bank score
Other: Questionnaire — assessment of emotional state using the Neuropathic Pain Symptom Inventory score (NPSI)
Other: Questionnaire — To assess whether pain measured by a Numercial rating scale (NRS) predicts chronic postoperative pain.

SUMMARY:
Sternotomy results in chronic postoperative pain in 30-55% of subjects. Few studies have been published on chronic pain in cardiac surgery, but there appears to be a relationship between the area of peri-scar hyperalgesia, which is indicative of postoperative hyperalgesia, and the occurrence of persistent pain 6 months after surgery. The aim of this study was therefore to assess whether the area of the postoperative hyperalgesia zone predicts chronic pain at 3 months post-surgery in cardiac surgery. To define the area of hyperalgesia at Day 2, pain mapping (algocartography) will be performed in patients who have had a sternotomy in cardiac surgery, together with pain assessment using the Simple Digital Pain Scale. Von Frey filaments of different sizes will be used for mapping. At Day 90, additional quality-of-life questionnaires will be carried out to check whether chronic pain is still present. A simple numerical scale (ENS) assessment at rest and during activity, and a record of pain-relieving treatments related to the surgery will also be carried out during this call.

The investigators hypothesize that the area of the zone of hyperalgesia assessed at Day 2 predicts the occurrence of chronic pain at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled surgery
* Conventional cardiac surgery by sternotomy: valve repair or replacement, coronary, thoracic aortic or combined surgery
* Age over 18
* No opposition from patient
* Patient affiliated to a social security

Exclusion Criteria:

* Emergency surgery
* Patient refusal
* Redux surgery
* Patients under guardianship
* History of drug addiction
* Preoperative opioid treatment
* Morbid obesity (body mass index >30kg/m2)
* Pregnant or breast-feeding women
* Patients taking part in another clinical study likely to interfere with the results of the present study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study focuses on adult patients undergoing scheduled cardiac surgery via sternotomy.
  84 patients required for the study Only patients operated at Hopital Louis Pradel will be included
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate whether the area of postoperative hyperalgesia predicts chronic pain at 3 months postoperatively in cardiac surgery. | 2 days after surgery
  To define the zone of hyperalgesia on Day 2, pain mapping will be carried out in patients who had a sternotomy in cardiac surgery. To this end, Von Frey filaments of different calibers will be used. Depending on the filament used and the discomfort or pain felt in different areas, we can construct a pain intensity map (or algocartography). To define chronic pain, we will use the NRS (Numerical Rating Scale) to measure pain. The gold standard is the occurrence of chronic postoperative pain defined by NRS > 3
Evaluate whether the area of postoperative hyperalgesia predicts chronic pain at 3 months postoperatively in cardiac surgery | 90 days after surgery
  To define the zone of hyperalgesia on Day 2, pain mapping will be carried out in patients who had a sternotomy in cardiac surgery. To this end, Von Frey filaments of different calibers will be used. Depending on the filament used and the discomfort or pain felt in different areas, we can construct a pain intensity map (or algocartography). To define chronic pain, we will use the NRS (Numerical Rating Scale) to measure pain. The gold standard is the occurrence of chronic postoperative pain defined by NRS > 3

SECONDARY OUTCOMES:
Assess whether pain measured by a NRS predicts chronic postoperative pain. | 48 first hours after surgery
  AUC of the ability of pain intensity assessment by NRS in the immediate postoperative period (first 48 hours) to predict the occurrence of chronic postoperative pain, and correlation test.
assess whether total morphine consumption at 3 days predicts chronic postoperative pain | 48 hours after surgery
  AUC ROC of the capacity of cumulative morphine consumption at day 3 to predict the onset of chronic postoperative pain, and correlation test
Evaluate the relationship between the area of the zone of hyperalgesia by mapping the second day and postoperative morphine consumption 3 days after surgery | During 48 first hours after surgery
  AUC ROC of the area of hyperalgesia at day 2 (area of hyperalgesia) to predict postoperative morphine consumption and correlation test
Evaluate the area of the hyperalgesia zone by mapping 2 days after surgery to predict the use of analgesics at 3 months postoperatively | 2 days after surgery
  AUC ROC of hyperalgesia area capacity at day 2 (hyperalgesia area surface), to predict analgesic consumption at 3 months and correlation test.
assess the relationship between the area of hyperalgesia by mapping 2 days after surgery and sleep quality at 3 months postoperatively. | 2 days after surgey
  AUC ROC of hyperalgesia area capacity at day (hyperalgesia area surface), to predict sleep quality (PROMIS item BANK scale)
assess the relationship between the area of hyperalgesia by mapping 2 days after surgery and sleep quality at 3 months postoperatively. | 90 days after surgey
  AUC ROC of hyperalgesia area capacity at day (hyperalgesia area surface), to predict sleep quality (PROMIS item BANK scale)
Evaluate the area of the zone of hyperalgesia by mapping 2days after surgery to predict neuropathic pain at 3 months postoperatively | 2 days after surgey
  AUC ROC of hyperalgesia area capacity at day 2 (areas of high pain intensity and hyperalgesia area surface), to predict neuropathic pain (NPSI: neuropathic pain symptom inventory) and correlation test.
Evaluate the area of the zone of hyperalgesia by mapping 2days after surgery to predict neuropathic pain at 3 months postoperatively | 90 days after
  AUC ROC of hyperalgesia area capacity at day 2 (areas of high pain intensity and hyperalgesia area surface), to predict neuropathic pain (NPSI: neuropathic pain symptom inventory) and correlation test
Assessing whether preoperative anxiety predicts chronic postoperative pain | 1 to 2 days before surgey
  AUC ROC of the ability of preoperative anxiety to predict the occurrence of chronic postoperative pain, and correlation test.

CONTACTS AND LOCATIONS:
Overall Officials: Judit JORDANA BOFILL, PI-nurse, Principal Investigator — Service d'Anesthésie Réanimation Hôpital Louis Pradel, Groupement Hospitalier Est 28 av. du Doyen Lépine
Locations (1):
- Service Anesthésie réanimation Hôpital Louis Pradel, Groupement Hospitalier Est Adresse 28 av. de Doyen Lépine 69677 BRON Cedex, Bron, France, France

IPD SHARING:
Plan to Share IPD: No